CLINICAL TRIAL: NCT02909205
Title: Development and Evaluation of a Care Protocol for Caregivers and Parents of Children Recently Gastrostomised
Brief Title: a Care Protocol for Caregivers and Parents of Children Recently Gastrostomised
Acronym: Gastrostomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D21537
Record Dates: First submitted 2016-08-29; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-08

CONDITIONS: Gastrostomy
Keywords: child; gastrostomy; supportive care; educational program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Other): First phase : before training / sensitization / booklet delivery
  Interventions: Other: sensitization / educational program
- post intervention (Other): Second phase : after training / sensitization / booklet delivery
  Interventions: Other: training / sensitization program

INTERVENTIONS:
Other: sensitization / educational program — the intervention program was built based on the results of the pre-intervention phase survey, about the knowledge of caregivers and parents of children with gastrostomy about gastrostomy management. It consists in booklets for caregivers and parents of children. This booklet is the support of a specific training of carers and parents of children who have recently benefitted from a gastrostomy
  Arms: control
Other: training / sensitization program — diffusion of gastrostomy in-hospital care protocols, and booklets for families. These tools have been prepared by a pilot group of professional of the investigating centers.
  Arms: post intervention

SUMMARY:
The aim of the study is to improve care practice related to gastrostomy management. This a before-after study, aimed at evaluating knowledge of care givers, families and patients about gastrostomy management. The intervention includes 1) A training in a care protocol for hospital care givers, and 2) A booklet for patients, families, and outpatient care givers. The evaluation criterion is a questionnaire to assess knowledge of hospital care givers, patients, families, and outpatient care givers.

ELIGIBILITY:
Inclusion Criteria:

* parents and hospital care givers of children undergoing gastrostomy who accept to participate.

Exclusion Criteria:

* family unable to understand French language, caregiver who has previously answered to the study questionnaire

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Change from knowledge score | Between day 0 and day 5
  The anonymised questionnaires are identified by a number assigned to the selected case; they include items about global knowledge about gastrostomy, its day to day use, possible complications, and surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric VALLA, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No